CLINICAL TRIAL: NCT04215315
Title: Prevalence and Characteristics of Fractures in Preterm Infants Presenting to Accident and Emergency: A Retrospective Study.
Brief Title: Fracture In Preterm Infants Study (FIPIN Study)
Status: Completed | Type: Observational
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SCH-2086
Record Dates: First submitted 2018-04-23; First posted 2020-01-02 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Fractures, Bone
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Retrospective observation — Case note and imaging review

SUMMARY:
Children who are born early (pre-term infants) are at increased risk of fractures until the age of 2 years, due to their weak bones caused by several physiological, and environmental factors.There is however little information about the persistence of this increased risk of fractures in childhood. There is also lack of detail in the medical literature about the gestational age at birth of children presenting to hospitals with fractures, the nature of their fractures and the differences in fracture features, if any, between the preterm and term (infants born at 37 weeks and above) children. This information would be especially useful for doctors when deciding if a fracture with no other obvious explanation in a preterm child is caused by an accidental or inflicted injury.

This dilemma is complicated by reports that preterm children are more likely to be subjected to abuse as compared to term children. Furthermore, infants less than a year old are more likely to be abused, and this coincides with the time when preterm infants are most vulnerable. Hence it is important to collect information about the physical examination, chemical substances in their blood and x-ray features of fractures in preterm children. Also important to study is whether there are differences in how accidental and inflicted fractures present in term and preterm children, as certain findings in term children might not apply in the context of prematurity. Determining if preterm birth is a major cause for childhood fractures is also especially relevant to the medico legal profession. When there is a suspected inflicted fracture in an ex-preterm child, the outcome could depend on whether prematurity is an adequate explanation for fractures. We would like to collect, study and present detailed information on the differences in causes and patterns of accidental and inflicted fractures in both preterm and term children. This could lend support to medical opinions offered in medico legal proceedings in which child abuse is alleged in preterm infants.

DETAILED DESCRIPTION:
This is a retrospective study involving only data collection and no patient contact.

Data will be collected from both Sheffield Children's Hospital Accident and Emergency Department and Jessop Hospital. The coding office will be contacted for a list of children below the age of 2 presenting to SCH with a fracture from January 2005 to December 2015, and a list of children born in Jessop Hospital over the same time period. By comparing both lists and selecting the matching cohort, we will have a list of those children (below the age of 2, preterm or term) born in Jessop Hospital who presented to SCH with a fracture over the last 10 years. The clinical notes of these patients will be accessed electronically and through their clinical files.

Data collection

Jessop:

A consultant employed by Jessop hospital or with the appropriate HR arrangement with the Trust will retrieve numbers of all pre-term babies born between Jan 2005 and Dec 2014 from the Jessop database and collect the data.

SCH:

A named researcher will retrieve NHS numbers of all children( both term and pre-term) less than 2 years of age presenting with a fracture between Jan 2005 and Dec 2014 from Sheffield Children's Hospital Coding Office and collect the data.

The PI of the study will cross match both records and identify the common cohort and assign one patient study identification number for each NHS number which should be used across both sites.

A named researcher will collect data from both Sheffield Children's Hospital Accident and Emergency Department and Jessop Hospital as outlined above.

Statistical analysis will be performed using SPSS. Descriptive for age, sex, gestation, ethnicity, and diagnosis; Chi-square for categorical data, with the possibility of regression analysis on advice of a statistician.

ELIGIBILITY:
Inclusion Criteria:

* Children (both term and preterm)up to age of 2, who have had either accidental or inflicted fractures and are otherwise healthy.

Exclusion Criteria:

* Children who have sustained fractures from other causes (post-surgery, post-resuscitation, metabolic bone diseases) or have any significant metabolic bone condition or received any medication known to affect vitamin D metabolism 3 months before enrolment (oral glucocorticoids, anticonvulsants etc.)

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Using medical records
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Total number of fractures sustained by each child | 9 Months
  Number

SECONDARY OUTCOMES:
Pattern (distribution) of fractures in those with fracture(s) | 9 months
  Number per bone

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Childrens NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No